CLINICAL TRIAL: NCT06040879
Title: Postoperative Analgesia Outcomes Of Pericapsular Nerve Group Block (PENG Block) Combined With Lateral Femoral Cutaneous Nerve Block After Hip Replacement Surgery: A Randomized Controlled Study
Brief Title: PENG Block and Lateral Femoral Cutaneous Nerve Block For Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HMU09.2023
Record Dates: First submitted 2023-09-07; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: POSTOPERATIVE ANALGESIA
Keywords: Pericapsular Nerve Group Block; lateral femoral cutaneous nerve; multimodal analgesia; ultrasound-guided analgesia; patient-controlled analgesia

STUDY DESIGN:
Intervention Model Description: PCA group and PENG BLOCK group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG BLOCK (Experimental): receiving pain relief through PENG and LFCN block
  Interventions: Procedure: PERICAPSULAR NERVE GROUP BLOCK COMBINED WITH LATERAL FEMORAL CUTANEOUS NERVE BLOCK
- PCA (Active Comparator): receiving morphine PCA analgesia
  Interventions: Procedure: PERICAPSULAR NERVE GROUP BLOCK COMBINED WITH LATERAL FEMORAL CUTANEOUS NERVE BLOCK

INTERVENTIONS:
Procedure: PERICAPSULAR NERVE GROUP BLOCK COMBINED WITH LATERAL FEMORAL CUTANEOUS NERVE BLOCK — During and after the surgery, a group of patients received intravenous morphine analgesia via PCA (concentration 1mg/ml, bolus dose of 1mg, lock time 10 minutes, maximum dose 10mg/4 hours). The remaining group of patients receive pain relief by PENG block and LFCN block. In this group, the ultrasound probe was placed horizontally from the anterior superior iliac spine, and was moved along the femoral arc defining the pubic spine. Then, the transducer was rotated 45 degrees, moved parallel to the femoral arch identifying the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE) and inferior lumbosacral head. The ultrasound probe was moved lightly until the upper end of the femoral head was identified. Next, a 120 mm Tuohy 18G anesthetic needle was used under ultrasound guidance, which was moved lateral to medial in the plane between the ultrasound transducer and the superior tip of the femoral head. Then, 10 mL of ropivacaine 0.25% was injected through the anesthetic needle tip

SUMMARY:
Background: this study aimed to describe the pain relief outcomes after hip replacement surgery by continuous Pericapsular Nerve Group Block (PENG Block) in combination with lateral femoral cutaneous nerve (LFCN) block under the guidance of ultrasound.

Methods: patients who had hip surgery at E University hospital, Hanoi, Vietnam from August 2021 to August 2022 belonged to two groups: group of patients with pain relief with PENG block in combination with LFCN block (PENG BLOCK group) and group of patients with patient-controlled intravenous analgesia (PCA group). Outcomes regarding clinical and pain score from initiation of insertion or PCA insertion (H0) to after 72 hours (H72) were recorded.

DETAILED DESCRIPTION:
First, patients were explained about the study and asked to sign written informed consent if they agreed to participate in the study. Next, the patient was instructed to use the visual analogue scale (VAS) for pain score, as well as how to press the button to request pain relief. Then, a monitor was installed and operated to assess the clinical parameters (electrocardiogram, blood pressure, SpO2, arterial blood pressure, temperature). The patient was oxygenated 3-5 liters/minute and performed a peripheral intravenous line, with an 18G catheter, infused with 0.9% NaCl solution. Spinal anesthesia was administered with ropivacaine 0.5% and fentanyl.

During and after the surgery, a group of patients received intravenous morphine analgesia via PCA (concentration 1mg/ml, bolus dose of 1mg, lock time 10 minutes, maximum dose 10mg/4 hours). The remaining group of patients receive pain relief by PENG block and LFCN block. In this group, the ultrasound probe was placed horizontally from the anterior superior iliac spine, and was moved along the femoral arc defining the pubic spine. Then, the transducer was rotated 45 degrees, moved parallel to the femoral arch identifying the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE) and inferior lumbosacral head. The ultrasound probe was moved lightly until the upper end of the femoral head was identified. Next, a 120 mm Tuohy 18G anesthetic needle was used under ultrasound guidance, which was moved lateral to medial in the plane between the ultrasound transducer and the superior tip of the femoral head. Then, 10 mL of ropivacaine 0.25% was injected through the anesthetic needle tip.

Data were collected at different times including: before surgery, before anesthesia, during surgery and after surgery. The information was recorded in the medical record.

Preoperative data: the collected information included the general characteristics of the study patients including age, gender, weight, height, history of smoking/motion sickness, diagnosis, health classification according to ASA, liver and kidney function tests. With pre-anesthesia data, information was collected including pulse, blood pressure, respiratory rate, SpO2.

Intraoperative data: the information collected includes information about anesthesia and surgical procedure.

Post-operative data: the collected information includes blood test results (urea, creatinine, liver enzymes), pain score (Visual analogue scale - VAS - scale from 0 to 10, the higher the score, the higher the pain level. more), analgesic drugs consumption status, respiratory and circulatory changes, adverse events, and analgesic satisfaction. Time was recorded from initiation of catheterization or PCA insertion (H0) to after 72 hours (H72).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III.
* Patients had hip replacement surgery.

Exclusion Criteria:

* infection of the anesthetized area.
* coagulation disorders
* organs dysfunction
* allergy to anesthetics
* did not cooperate with physicians
* history of opioid dependence
* inability to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
VAS score at rest and on movement | Time was recorded from initiation of catheterization or PCA insertion (H0) to after 72 hours (H72)
  the average VAS score (Visual Analogue Scale) at rest and on movement of both groups. The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark.
Side effects | Time was recorded from initiation of catheterization or PCA insertion (H0) to after 72 hours (H72)
  Rate of vomitting/nausea, itchy, urinary retention, respiratory failure postoperative of both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tu Nguyen, Professor, Study Director — Hanoi Medical University
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
We agree that all results and conclusion of this research will be used fully for other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from September 2023 to the unidentified time
Access Criteria: anesthesiologists, surgeons all over the world

REFERENCES:
- [Result] Ferguson RJ, Palmer AJ, Taylor A, Porter ML, Malchau H, Glyn-Jones S. Hip replacement. Lancet. 2018 Nov 3;392(10158):1662-1671. doi: 10.1016/S0140-6736(18)31777-X. PMID 30496081
- [Result] Ferrata P, Carta S, Fortina M, Scipio D, Riva A, Di Giacinto S. Painful hip arthroplasty: definition. Clin Cases Miner Bone Metab. 2011 May;8(2):19-22. PMID 22461810
- [Result] YaDeau JT, Tedore T, Goytizolo EA, Kim DH, Green DS, Westrick A, Fan R, Rade MC, Ranawat AS, Coleman SH, Kelly BT. Lumbar plexus blockade reduces pain after hip arthroscopy: a prospective randomized controlled trial. Anesth Analg. 2012 Oct;115(4):968-72. doi: 10.1213/ANE.0b013e318265bacd. Epub 2012 Jul 19. PMID 22822195
- [Result] Duarte LT, Beraldo PS, Saraiva RA. [Effects of epidural analgesia and continuous lumbar plexus block on functional rehabilitation after total hip arthroplasty]. Rev Bras Anestesiol. 2009 Sep-Oct;59(5):531-44. doi: 10.1016/s0034-7094(09)70078-9. Portuguese. PMID 19784509
- [Result] Singelyn FJ, Ferrant T, Malisse MF, Joris D. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous femoral nerve sheath block on rehabilitation after unilateral total-hip arthroplasty. Reg Anesth Pain Med. 2005 Sep-Oct;30(5):452-7. doi: 10.1016/j.rapm.2005.05.008. PMID 16135349
- [Result] Lin DY, Morrison C, Brown B, Saies AA, Pawar R, Vermeulen M, Anderson SR, Lee TS, Doornberg J, Kroon HM, Jaarsma RL. Pericapsular nerve group (PENG) block provides improved short-term analgesia compared with the femoral nerve block in hip fracture surgery: a single-center double-blinded randomized comparative trial. Reg Anesth Pain Med. 2021 May;46(5):398-403. doi: 10.1136/rapm-2020-102315. Epub 2021 Feb 26. PMID 33637625
- [Result] Shafiq F, Hamid M, Samad K. Complications and interventions associated with epidural analgesia for postoperative pain relief in a tertiary care hospital. Middle East J Anaesthesiol. 2010 Oct;20(6):827-32. PMID 21526668
- [Result] Rasouli MR, Viscusi ER. Adductor Canal Block for Knee Surgeries: An Emerging Analgesic Technique. Arch Bone Jt Surg. 2017 May;5(3):131-132. No abstract available. PMID 28656158
- [Result] Kamel I, Ahmed MF, Sethi A. Regional anesthesia for orthopedic procedures: What orthopedic surgeons need to know. World J Orthop. 2022 Jan 18;13(1):11-35. doi: 10.5312/wjo.v13.i1.11. eCollection 2022 Jan 18. PMID 35096534
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/musculoskeletal-conditions